CLINICAL TRIAL: NCT01779973
Title: Remote Observed Dosing to Increase Suboxone Compliance
Acronym: RODISC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 816651
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-04

CONDITIONS: Opiate Dependence
Keywords: Skype; compliance; remote dosing; suboxone; opiate; opiates; heroin; oxycontin; Philadelphia
MeSH Terms: conditions — Opioid-Related Disorders; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Remote Observed Dosing (Experimental): Compliance with dosage observations of suboxone doses using remote observed dosing 4 days per week and 1 weekly in-office visit.
  Interventions: Behavioral: Remote Observed Dosing

INTERVENTIONS:
Behavioral: Remote Observed Dosing

SUMMARY:
The goal of this project is to test the feasibility, acceptability, and preliminary efficacy of using remote compliance monitoring in buprenorphine (Suboxone®) treatment for opiate dependence. To that end, 10 opiate dependent subjects will be recruited through the University of Pennsylvania's Treatment Research Center, an outpatient substance abuse treatment facility. All subjects will receive buprenorphine (Suboxone®) (16 mg/day, adjusted as needed according to individual requirements).

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily provide written informed consent prior to the conduct of any study-related procedure
* Male or female, 18 to 65 years of age,
* Meet DSM-IV criteria for current opioid dependence
* Females of childbearing potential and fertile males must use a reliable means of contraception
* Owns a smartphone with forward facing camera that allows for use of Skype

Exclusion Criteria:

* University of Pennsylvania student, employee, or affiliate
* Current diagnosis of AIDS
* Presence of AST and/or ALT equal to or 3X upper limit of normal
* Total bilirubin and/or creatinine equal to or 1.5X upper limit or normal
* Current diagnosis of chronic pain requiring opioids
* Pregnant or lactating females
* Previous hypersensitivity or allergy to buprenorphine or EVA-containing substances
* Current use of agents metabolized through CYP 3A4 such as azole antifungals (e.g. ketoconazole), macrolide antibiotics (e.g. erythromycin), and protease inhibitors (e.g. ritonavir, indinavir, saquinavir)
* Meet DSM-IV criteria for current dependence on any psychoactive substances other than opioids or nicotine (e.g. alcohol, sedatives)
* Current use of benzodiazepines other than physician prescribed
* Significant medical or psychiatric symptoms or dementia which in the opinion of the investigators would preclude compliance with the protocol, adequate cooperation in the study, or obtaining informed consent
* Concurrent medical conditions (such as severe respiratory insufficiency) that may prevent the patient from safely participating in the study; and/or any pending legal action that could prohibit participation and/or compliance in study procedures
* Participated in a clinical study within the previous 8 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The number of suboxone dose taken during the course of the study. The number of opiate-negative urine samples provided during the study. | 9 months

SECONDARY OUTCOMES:
Patterns of missed doses including visit times and frequency impact. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer G Plebani, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States